CLINICAL TRIAL: NCT04831320
Title: Nab-Paclitaxel in Combination With Nivolumab to Treat Recurrent or Metastatic Head and Neck Squamous-Cell Carcinoma That Progressed on a PD-1 or PD-L1 Inhibitor: A Single-Arm, Phase 2 Trial
Brief Title: Nab-Paclitaxel in Combination With Nivolumab to Treat Recurrent or Metastatic Head and Neck Squamous-Cell Carcinoma That Progressed on a PD-1 or PD-L1 Inhibitor
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202105128
Record Dates: First submitted 2021-03-31; First posted 2021-04-05 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Head-and-neck Squamous-cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- nab-Paclitaxel + Nivolumab (Experimental): * nab-Paclitaxel 125 mg/m^2 intravenous (IV) on days 1, 8 & 15 of each 28-day cycle.
  * Nivolumab 480 mg IV Day 1 of each 28-day cycle.
  Interventions: Drug: nab-paclitaxel; Drug: Nivolumab

INTERVENTIONS:
Drug: nab-paclitaxel — Supplied by Celgene Corporation
  Other Names: Abraxane
Drug: Nivolumab — Supplied by Bristol-Myers Squibb
  Other Names: Opdivo

SUMMARY:
The primary hypothesis is that the objective response rate (ORR) with nab-paclitaxel and nivolumab will be significantly higher than the historical control (ORR 30%).

The KEY secondary hypothesis is that the median PFS with nab-paclitaxel and nivolumab will be significantly longer than the historical control (median PFS 3.6 months).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed recurrent or metastatic HNSCC of the oral cavity, larynx, hypopharynx, oropharynx, or p16 positive neck node with unknown primary (but clinically thought to be oropharynx).
* Known p16 status (positive or negative) if oropharynx or unknown primary of the neck.
* Measurable disease per RECIST. Measurable disease defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 10 mm with CT scan, as ≥ 20 mm by chest x-ray, or ≥ 10 mm with calipers by clinical exam.
* Progression of disease, as assessed by RECIST, that occurred on a PD-1 or PD-L1 inhibitor (given alone or with other therapy) to treat recurrent or metastatic disease. Progression of disease that occurred on a PD-1 or PD-L1 inhibitor given as a component of a curative-intent regimen is excluded.
* PD-L1 CPS by IHC (22C3 antibody) on tumor tissue is strongly encouraged to be available or performed, although the test result is not required to enroll onto the trial. Patients with tumor PD-L1 TPS (but not CPS) available are also eligible; but, PD-L1 CPS should be performed in these cases. Fresh tumor tissue (obtained after progression on prior PD-1 or PD-L1 inhibitor given for recurrent or metastatic disease) is strongly preferred, but archived tumor tissue from recurrence or initial diagnosis is also acceptable.
* At least 18 years of age.
* ECOG performance status < 1
* Normal bone marrow and organ function as defined below:

  * Hemoglobin > 9 g/L
  * Absolute neutrophil count ≥ 1,500/mcl
  * Platelets ≥ 100,000/mcl (transfusion independent, defined as not receiving platelet transfusions within 7 days prior to laboratory sample)
  * Total bilirubin ≤ 1.5 mg/dL
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 x IULN (in cases of bone mets or liver mets, AST/ALT < 5 x IULN)
  * Serum creatinine <1.5 x IULN or creatinine clearance > 50 mL/min by Cockcroft-Gault
* The effects of nivolumab and nab-paclitaxel on the developing human fetus are unknown. For this reason and because monoclonal antibodies and antimicrotubule agents are known to be teratogenic, women of childbearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry, for the duration of study participation, and for 6 months after the last dose of study treatment. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable) before the performance of any protocol-related procedures.

Exclusion Criteria:

* A history of other malignancy with the exception of malignancies for which all treatment was completed at least 1 year before registration and the patient has no evidence of disease.
* Has known active CNS metastases. Subjects with previously treated brain metastases may participate provided they are stable (without any evidence of progression by imaging 4 weeks prior to the first dose of study treatment and any neurologic symptoms have stabilized), have no evidence of new or enlarging brain metastases, and are on stable or tapering doses of steroids for at least 14 days prior to first dose of study treatment.
* A history of serious allergic reactions attributed to compounds of similar chemical or biologic composition to agents used in the study (Allergic reaction to cetuximab is allowed as there are other standard of care options for the investigator's choice arm).
* Receiving systemic corticosteroid therapy (in doses exceeding 10 mg daily of prednisone equivalent) within 7 days prior to the first dose of treatment. A history of severe autoimmune disorder requiring high-dose corticosteroid treatment due to prior PD-1 inhibitor is an exclusion criterion.
* Greater than Grade 2 pre-existing peripheral neuropathy (per CTCAE).
* Uncontrolled serious intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative serum pregnancy test within 24 hours prior to the start of study treatment.
* Prior organ or allogeneic stem cell transplant.
* Has an active autoimmune disease (i.e. rheumatoid arthritis, lupus, Sjogren's syndrome) that has required IV or subcutaneous systemic treatment in the past 6 months (excluding Rituxan). Replacement therapy (i.e. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Prisoners, or subjects who are compulsory detained.
* Prior taxane (including paclitaxel or docetaxel) given to treat recurrent or metastatic disease.
* Prior taxane (including paclitaxel or docetaxel) given as a component of a curatively intended multimodality therapy IF the latter was completed within 6 months of subsequent development of recurrent or metastatic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) as assessed by RECIST 1.1 | Through completion of treatment (estimated to be 4 months)
  * ORR: Proportion of patients who achieve a complete or partial response to treatment
  * Complete Response (CR): Disappearance of all target lesions. Disappearance of all non-target lesions and normalization of tumor marker level. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  * Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Through completion of follow-up (estimated to be 13 months)
  * PFS, defined as the days from the date of treatment to the first documentation of disease progression or death from any cause, whichever occurs first. The alive patients without progression are censored at the date of last follow-up. The patients without progression will not receive anti-cancer therapy, but the patients who have progression may receive additional anti-cancer therapy.
  * Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Duration of response (DOR) | Through completion of treatment (estimated to be 4 months)
  * Duration of overall response: The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started).
  * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Disappearance of all non-target lesions and normalization of tumor marker level.
  * Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Incidence of adverse events | Through 100 days after completion of treatment (estimated to be 7.5 months)
Incidence of immune-related adverse events | Through 100 days after completion of treatment (estimated to be 7.5 months)
Number of dose reductions of nab-paclitaxel | Through completion of treatment (estimated to be 4 months)
Number of dose reductions of nivolumab | Through completion of treatment (estimated to be 4 months)
Number of dose delays of nab-paclitaxel | Through completion of treatment (estimated to be 4 months)
Number of dose delays of nivolumab | Through completion of treatment (estimated to be 4 months)
Number of dose interruptions of nab-paclitaxel | Through completion of treatment (estimated to be 4 months)
Number of dose interruptions of nivolumab | Through completion of treatment (estimated to be 4 months)
Overall survival (OS) | Through completion of follow-up (estimated to be 13 months)
  -OS: defined as the days from the date of treatment to death from any cause, censored at the date of last follow-up otherwise.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas R Adkins, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu